CLINICAL TRIAL: NCT03947294
Title: Clinical Evaluation of the Ease of Use of a New Indirect Calorimeter in Canopy and Face Mask Modes for Energy Expenditure Measurement: The ICALIC 2 International Multicentric Study (Second Phase)
Brief Title: The ICALIC 2 International Multicentric Study
Acronym: ICALIC2
Status: Terminated | Type: Observational
Why Stopped: No participation of centers outside Switzerland because of difficulty in recruiting during a Covid pandemic.
Sponsor: Prof. Claude Pichard (Other)
Responsible Party: Sponsor-Investigator, Prof. Claude Pichard, Head, Clinical Nutrition, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2019-00106
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Cancer; Surgery; Hemodialysis
Keywords: Indirect calorimetry; Energy expenditure; VO2; VCO2
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Q-NRG® — Energy expenditure measurements
  Other Names: Currently used calorimeters

SUMMARY:
Clinicians need to measure energy expenditure (EE) by indirect calorimetry (IC) to optimize nutritional support for a better clinical outcome, especially in patients with chronic conditions or with high risk of under- and over- feeding. However, IC is rarely used in clinical routine because the devices currently on the market are of tedious use, imprecise and expensive. An easy-to-use, accurate and inexpensive IC device (Q-NRG® CE marking n°MED 9811) has been developed to meet specifications made by and for clinicians. The ease of use of this new IC device has been first evaluated in mechanical ventilation mode. This second phase aims at evaluating the ease of use, the stability and the feasibility of the measurements with this new IC device in canopy and face mask modes for spontaneously breathing adult patients.

DETAILED DESCRIPTION:
This study aims at evaluating the ease of use, the stability and the feasibility of EE measurements with the new IC device in spontaneously breathing adult patients with malnutrition, cancer, surgery or haemodialysis, using the canopy and face mask modes.

Patient data will be obtained from the medical records before EE measurement. EE measurement will be performed sequentially with the Q-NRG® and the IC device currently used in each study center. Patient data input, calibration, installation of face mask or canopy hood on the patient, and EE measurement recording will be performed according to the procedure stated in their respective user manual. Time needed to perform EE will be calculated afterwards from the time the IC device is turned on to EE measurement reaches a steady state with a variation ≤10%.

In a subset of 15 subjects, accuracy of gas composition (O2 and CO2) measurement by the Q-NRG® will be assessed by comparison with the reference method consisting in a mass spectrometer.

ELIGIBILITY:
Inclusion Criteria:

All spontaneously breathing adult patients (≥ 18 years) referred to the Nutrition Unit in the context of malnutrition, cancer, surgery or haemodialysis.

Exclusion Criteria:

1. < 18 years
2. Intolerance or phobia to canopy or face mask
3. Physical agitation or activity (< 1hr before EE measurement)
4. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spontaneously breathing adult patients with malnutrition, cancer, surgery or haemodialysis.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Time needed to perform EE measurement. | Immediately after the measurement
  Time needed to perform EE will be calculated from the time the Q-NRG® or the currently used calorimeter is turned on to EE measurement reaches a steady state with a variation ≤10%.

SECONDARY OUTCOMES:
Accuracy and precision of VO2, VCO2, RQ and EE measurements. | Immediately after the measurement.
  Accuracy and precision of VO2, VCO2, RQ and EE measurements with the Q-NRG® in face mask or canopy mode will be compared to currently used indirect calorimeters.
Coefficient of variation of VO2, VCO2, RQ and EE. | Immediately after the measurement.
  The stability of VO2, VCO2, RQ and EE measurements with the Q-NRG® in face mask or canopy mode will be compared to currently used indirect calorimeters.
Clinical condition restriction. | Immediately after the measurement.
  Clinical conditions, if any, precluding or disturbing the EE measurement with the Q-NRG®.

OTHER OUTCOMES:
Accuracy of O2 and CO2 analysis. | Immediately after the measurement.
  Accuracy of gas composition (O2 and CO2) measurement by the Q-NRG® assessed by comparison with a mass spectrometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Geneva 14, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupertuis YM, Delsoglio M, Hamilton-James K, Berger MM, Pichard C, Collet TH, Genton L. Clinical evaluation of the new indirect calorimeter in canopy and face mask mode for energy expenditure measurement in spontaneously breathing patients. Clin Nutr. 2022 Jul;41(7):1591-1599. doi: 10.1016/j.clnu.2022.05.018. Epub 2022 May 27. PMID 35671611